CLINICAL TRIAL: NCT02849652
Title: Testing an Organizational Change Model to Address Smoking in Mental Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823871; R01CA202699 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-29 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Nicotine Dependence
Keywords: Smoking cessation; Nicotine dependence; Organizational change; Mental Healthcare
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATTOC (Experimental): Addressing Tobacco Through Organizational Change is a multi-phase organizational intervention to promote the treatment of tobacco dependence
  Interventions: Behavioral: ATTOC Intervention
- Usual Care (Other): Usual Care is the typical guideline based smoking cessation intervention
  Interventions: Behavioral: UC Intervention

INTERVENTIONS:
Behavioral: ATTOC Intervention — ATTOC is implemented in a systematic 3-phase process with 10 steps to guide sites through cultural change and implementation of evidence-based practice.
  Arms: ATTOC
Behavioral: UC Intervention — Sites randomized to UC will not receive an organizational intervention to address TUD treatment. To ensure standardization across UC sites, study personnel will provide a 1-day training seminar that will include written materials describing recommended treatments for TUD to UC personnel consistent with established treatment guidelines.
  Arms: Usual Care

SUMMARY:
Despite an overall reduction in US smoking rates from >50% in the 1960s to about 20% by 2000, the rate of smoking among persons with a serious mental illness (SMI) remains 2-3 times greater than in the general population. Further, even the recent small decline in smoking rates that has been reported in the general population in the past decade has not occurred among smokers with an SMI. In fact, 44% of all the cigarettes consumed in the US are by individuals with a psychiatric disorder and the primary cause of death among Americans with an SMI is a tobacco-related disease.

This cluster randomized trial will be conducted in 14 Philadelphia community mental health clinics (CMHCs). Clinics will be randomized to either Addressing Tobacco Through Organizational Change model (ATTOC) or Usual Care (UC) treatment groups. The investigators hypothesize that 1) at the end of the intervention and at a 3-month follow-up, rates of adherence to guidelines for treating TUD will be greater among clinic personnel that receive the ATTOC intervention vs. clinic personnel in usual care; 2) at the end of the intervention and at a 3-month follow-up, rates of client smoking cessation will be significantly greater in clinics that receive the ATTOC intervention than among clients treated with usual care; and 3) using non-inferiority testing, at the end of the intervention and at a 3-month follow-up, there will be no significant degradation in mental health functioning or QOL among clients who receive care at clinics that received the ATTOC intervention than among clients treated with usual care.

DETAILED DESCRIPTION:
Despite an overall reduction in US smoking rates from >50% in the 1960s to about 20% by 2000, the rate of smoking among persons with a serious mental illness (SMI) remains 2-3 times greater than in the general population. Transforming the mental healthcare system to integrate and adhere to evidence-based guidelines for the provision of tobacco use disorder (TUD) treatment is a priority of the National Institute of Mental Health and is a critical component of a national effort to meet Healthy People 2020 target goals for tobacco use (www.healthypeople.gov).

The Addressing Tobacco Through Organizational Change (ATTOC) model is a systems-level intervention to address systemic and cultural barriers that undermine assessment and treatment of TUD. In this innovative way, ATTOC assumes that effective organizational change requires more than clinic personnel training; it also requires the application of organizational theory to address attitudinal and system barriers and promote a culture in which tobacco use is not accepted or supported and that TUD treatment is integrated into standard practice. Consistent with organizational theory, ATTOC is implemented in 3 phases: preparing for, implementing, and sustaining change. By addressing cultural barriers and strengthening the care system (e.g., integrated treatment), ATTOC intends to have sustained benefits beyond the intervention.

This cluster-randomized trial will be conducted with 14 Philadelphia CMHCs, 7 randomized to ATTOC and 7 to usual care (UC). Following randomization, study staff will visit sites to recruit clinic personnel and clients over a 4 to 6 week period. Those eligible will complete informed consent and HIPAA forms and a baseline assessment to establish pre-intervention levels on all measures (baseline). After 4-6 weeks, the ATTOC intervention will be implemented over 9 months, from Week 1 to Week 36 (with UC at the control sites). Two mid-intervention assessments (Weeks 12 and 24) will allow for performance feedback and mediational analyses. Week 36 (end-of-treatment; EOT) and 52 (3-months post-EOT) assessments will allow for evaluation of changes on outcomes between groups over time. All measures will be conducted at the respective CMHC (or over the phone if necessary) and 7-day point prevalence smoking cessation will be verified using a breath carbon monoxide (CO) monitor (abstinence = < 8ppm).

This will be the first controlled, randomized trial to evaluate the effects of the ATTOC model on clinician adherence to treatment guidelines, client smoking, and client mental health and QOL. If this approach is shown to be effective and safe, it can serve as a model for the nation's community mental healthcare infrastructure, representing a powerful initiative to address tobacco use in an under-served sub-group of smokers, and support efforts to attain the Healthy People 2020 goals regarding tobacco use.

ELIGIBILITY:
Inclusion Criteria (clinic client participants):

* Must be a client at a participating community mental health clinic
* Must be 18 years of age or older
* Must report daily average smoking of 5 cigarettes/day for the past 6 months
* Must have a documented Diagnostic and Statistical Manual Axis I or II disorder
* Must demonstrate the ability to communicate in English and provide written informed consent

Exclusion Criteria (clinic client participants):

* Exclusive use of electronic cigarettes (dual use with standard cigarettes will not be exclusionary)

Inclusion Criteria (Clinic personnel participants):

* Must be 18 years of age or older
* Must perform clinical care or supervisory duties
* Must demonstrate the ability to communicate in English and provide written informed consent

Exclusion Criteria:

* no clinical responsibilities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2016-07; Primary Completion 2022-08 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the final analyses are conducted to address the specific aims of this project, study data will be made available to other qualified researchers. The investigators plan to create a mechanism to allow such researchers to apply for access to these data.
Supporting Information: Study Protocol, ICF
Time Frame: Final analyses will be conducted after all participant activities have been completed, approximately 9/2021. Once the final analyses are conducted to address the specific aims of this project, study data will be made available.
Access Criteria: Study data will be made available to other qualified researchers. The investigators plan to create a mechanism to allow such researchers to apply for access to these data.

RESULTS

PARTICIPANT FLOW:
Groups:
- ATTOC Clients: Addressing Tobacco Through Organizational Change is a multi-phase organizational intervention to promote the treatment of tobacco dependence
  ATTOC Intervention: ATTOC is implemented in a systematic 3-phase process with 10 steps to guide sites through cultural change and implementation of evidence-based practice.
- ATTOC Staff: Addressing Tobacco Through Organizational Change is a multi-phase organizational intervention to promote the treatment of tobacco dependence
  ATTOC Intervention: ATTOC is implemented in a systematic 3-phase process with 10 steps to guide sites through cultural change and implementation of evidence-based practice.
  Staff from community mental healthcare clinics.
- Usual Care Clients: Usual Care is the typical guideline based smoking cessation intervention
  UC Intervention: Sites randomized to UC will not receive an organizational intervention to address TUD treatment. To ensure standardization across UC sites, study personnel will provide a 1-day training seminar that will include written materials describing recommended treatments for TUD to UC personnel consistent with established treatment guidelines.
- UC Staff: Usual Care is the typical guideline based smoking cessation intervention
  UC Intervention: Sites randomized to UC will not receive an organizational intervention to address TUD treatment. To ensure standardization across UC sites, study personnel will provide a 1-day training seminar that will include written materials describing recommended treatments for TUD to UC personnel consistent with established treatment guidelines.
  Staff from community mental healthcare clinics.
Period: Overall Study
Arm/Group | ATTOC Clients | ATTOC Staff | Usual Care Clients | UC Staff
Started | 344 | 131 | 266 | 91
Week 12 | 294 | 120 | 222 | 78
Week 24 | 279 | 112 | 188 | 74
Week 36 | 250 | 104 | 166 | 66
Week 52 | 230 | 94 | 142 | 65
Completed | 230 | 94 | 142 | 65
Not Completed | 114 | 37 | 124 | 26
Not completed — Lost to Follow-up | 104 | 35 | 116 | 22
Not completed — Withdrawal by Subject | 10 | 2 | 8 | 4

BASELINE CHARACTERISTICS:
Population: Descriptive statistics characterized the sample; chi-square for categorical variables (e.g., race) and ANOVA for continuous variables (e.g., age) compared the study arms. Variables that were significantly different across arms were included as covariates in modeling of outcomes.
Groups:
- Usual Care Staff: Usual Care is the typical guideline based smoking cessation intervention
  UC Intervention: Sites randomized to UC will not receive an organizational intervention to address TUD treatment. To ensure standardization across UC sites, study personnel will provide a 1-day training seminar that will include written materials describing recommended treatments for TUD to UC personnel consistent with established treatment guidelines.
- ATTOC Staff: Addressing Tobacco Through Organizational Change is a multi-phase organizational intervention to promote the treatment of tobacco dependence
  ATTOC Intervention: ATTOC is implemented in a systematic 3-phase process with 10 steps to guide sites through cultural change and implementation of evidence-based practice.
- Total: Total of all reporting groups
Arm/Group | Usual Care Clients | ATTOC Clients | Usual Care Staff | ATTOC Staff | Total
Number analyzed (Participants) | 266 | 344 | 91 | 131 | 832
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 266 | 344 | 91 | 131 | 832
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.8) | 48.3 (11.8) | 38.8 (15.6) | 45.5 (13.4) | 44.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 140 | 75 | 99 | 445
  Male | 135 | 204 | 16 | 32 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 31 | 9 | 8 | 84
  Not Hispanic or Latino | 222 | 306 | 70 | 93 | 691
  Unknown or Not Reported | 8 | 7 | 12 | 30 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 1 | 5
  Asian | 2 | 2 | 8 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 152 | 205 | 33 | 77 | 467
  White | 78 | 103 | 41 | 42 | 264
  More than one race | 6 | 15 | 4 | 3 | 28
  Unknown or Not Reported | 27 | 16 | 4 | 7 | 54
Region of Enrollment [Number; unit: participants]
  United States | 266 | 344 | 91 | 131 | 832

OUTCOME MEASURES:

1. Primary Outcome: Client Reported Tobacco Medications
Description: Client-reported use of tobacco treatment for nicotine dependence measured via self-report
Time Frame: Week 36 & Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Participants
  Week 36 | 48 | 28
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 62 | 24

2. Primary Outcome: Rate of Medication to Treat Nicotine Dependence - EHR
Description: Frequency of provision of medications for nicotine dependence measured via electronic health record (EHR) data for clients.
Time Frame: Week 36 & Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Participants
  Week 36 | 20 | 33
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 20 | 21

3. Secondary Outcome: Smoking Cessation Rate
Description: Change in proportion of smoking from baseline to follow-up time-points for clients
Time Frame: Week 36 & Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Participants
  Week 36 | 11 | 4
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 17 | 9

4. Secondary Outcome: Mental Health Functioning
Description: Mental health functioning was measured using the Revised Behavior and Symptom Identification Scale (BASIS-R), a 24-item assessment of mental health functioning that yields a total score and subscale scores for: depression, interpersonal relationships, self-harm, emotional liability, psychosis, and substance abuse. The total overall score was used. The 24 questions are scored on a 5-pointscale (from 0 to 4) with higher numbers indicating greater symptom/problem frequency or severity. The overall score can range from a 0 to a 96.
Time Frame: Week 36 & Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Scores on a scale
  Week 36 | 27.3 (21.5) | 31.8 (24.4)
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 28.7 (23.6) | 30.9 (25.0)

5. Secondary Outcome: Short-Form Health Survey Emotional
Description: The SF-12 (short form health survey) is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. For this outcome, the summed scores are from the emotional section of questionnaire. Higher scores signify lower QOL (quality of life) and the range of scores is 8-30.
Time Frame: Week 36 & Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from SF-12 (emotion questions)
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Score from SF-12 (emotion questions)
  Week 36 | 18.6 (3.8) | 18.5 (4.3)
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 17.9 (4.2) | 18.8 (4)

6. Secondary Outcome: Short-Form Health Survey Physical
Description: The SF-12 (short form health survey) is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. For this outcome, the summed scores are from the physical functioning section of the questionnaire. Higher scores signify lower QOL (quality of life) and the range of scores is 5-15.
Time Frame: Week 36 and Week 52
Population: Below is it specified the number of participants were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from SF-12 (physical questions)
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Score from SF-12 (physical questions)
  Week 36 | 9.5 (2.8) | 9.8 (2.9)
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 9.6 (2.7) | 10.1 (2.7)

7. Other Pre Specified Outcome: S-KAP: Staff-Reported Tobacco Treatment Treatment
Description: The Smoking Knowledge, Attitudes, and Practices instrument is composed of 5 scales that assess system and cultural barriers to providing treatment for smoking (from the healthcare provider perspective). The scores are from the summed items. Higher scores equal more tobacco treatment and the range of scores is 0-26.
Time Frame: Week 36 and Week 52
Population: Below it is specified the number of participants that were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from S-KAP
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 104 | 66
Score from S-KAP
  Week 36 | 12.3 (8.1) | 10.2 (7)
  Week 52: number analyzed (Participants) | 94 | 65
  Week 52 | 12.8 (8.6) | 11.6 (7.4)

8. Other Pre Specified Outcome: S-KAP: Staff-Reported Barriers to Treat Tobacco
Description: The Smoking Knowledge, Attitudes, and Practices instrument is composed of 5 scales that assess system and cultural barriers to providing treatment for smoking (from the healthcare provider perspective). The scores are from the summed items. Higher scores equal more barriers to tobacco treatment with the range of scores being 0-13.
Time Frame: Week 36 and Week 52
Population: Below it is specified the number of participants that were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from S-KAP
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 104 | 66
Score from S-KAP
  Week 36 | 11.5 (4.5) | 8.1 (2.5)
  Week 52: number analyzed (Participants) | 94 | 65
  Week 52 | 11.6 (4.6) | 7.7 (2.6)

9. Other Pre Specified Outcome: S-KAS: Client Reported Tobacco Treatment Treatment From Staff
Description: The Smoking Knowledge, Attitudes, and Services (S-KAS) survey assesses barriers to treating nicotine dependence from the client's perspective. The scores are from the summed items. Higher scores mean more tobacco treatment and the range of scores is 7-35.
Time Frame: Week 36 and Week 52
Population: Below it is specified the number of participants that were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from S-KAS
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Score from S-KAS
  Week 36 | 16.7 (6.2) | 15.9 (5.9)
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 16.3 (6.5) | 15.5 (6)

10. Other Pre Specified Outcome: S-KAP: Staff-Reported Skills to Treat Tobacco Treat Tobacco
Description: The Smoking Knowledge, Attitudes, and Practices instrument is composed of 5 scales that assess system and cultural barriers to providing treatment for smoking (from the healthcare provider perspective).The scores are from the summed items. Higher scores equal more skills and the range of scores is: 0-26.
Time Frame: Week 36 and Week 52
Population: Below it is specified the number of participants that were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from S-KAP
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 104 | 66
Score from S-KAP
  Week 36 | 14 (2.6) | 12.9 (3)
  Week 52: number analyzed (Participants) | 94 | 65
  Week 52 | 14 (2.7) | 13.5 (2.6)

11. Other Pre Specified Outcome: S-KAS: Client Reported Tobacco Services and Policies Services and Policies
Description: The Smoking Knowledge, Attitudes, and Services (S-KAS) survey assesses barriers to treating nicotine dependence from the client's perspective. The scores are from the summed items Higher scores equal more tobacco services. The range of scores is: 1-14.
Time Frame: Week 36 and Week 52
Population: Below it is specified the number of participants that were analyzed at each timepoint for this outcome
Measure: Mean (Standard Deviation); unit: Score from S-KAS
Arm/Group | ATTOC | Usual Care
Number analyzed (Participants) | 250 | 166
Score from S-KAS
  Week 36 | 6.8 (3.6) | 5.5 (3.2)
  Week 52: number analyzed (Participants) | 230 | 142
  Week 52 | 6.5 (3.5) | 5.6 (3.6)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at their week 36 and week 52 visit. Adverse events were monitored through from enrollment through study completion, up to 60 weeks.
Description: The definition of an adverse event matches the clinicaltrials.gov definition.
Groups:
- ATTOC Personnel: Addressing Tobacco Through Organizational Change is a multi-phase organizational intervention to promote the treatment of tobacco dependence
  ATTOC Intervention: ATTOC is implemented in a systematic 3-phase process with 10 steps to guide sites through cultural change and implementation of evidence-based practice.
  Staff from community mental healthcare clinics.
- Usual Care Personnel: Usual Care is the typical guideline based smoking cessation intervention
  UC Intervention: Sites randomized to UC will not receive an organizational intervention to address TUD treatment. To ensure standardization across UC sites, study personnel will provide a 1-day training seminar that will include written materials describing recommended treatments for TUD to UC personnel consistent with established treatment guidelines.
  Staff from community mental healthcare clinics.
Arm/Group | ATTOC Clients | Usual Care Clients | ATTOC Personnel | Usual Care Personnel
All-Cause Mortality (participants affected / at risk) | 8/344 | 6/266 | 2/131 | 0/91
Serious Adverse Events (participants affected / at risk) | 34/344 | 15/266 | 0/131 | 0/91
Other Adverse Events (participants affected / at risk) | 0/344 | 0/266 | 0/131 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATTOC Clients (N=344) | Usual Care Clients (N=266) | ATTOC Personnel (N=131) | Usual Care Personnel (N=91)
ORG0010 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 3/15/2017, ORG0010 was reportedly hospitalized for a duration of 30 days due to a psychotic episode and hearing voices. We were informed of this information from the participant on 6/5/2017, during their Week 36 visit.
ORG0008 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 4/13/2017, ORG0008 was reportedly hospitalized for a duration of 5 days due to a psychotic episode. We were informed of this information from the participant on 6/8/2017, during their Week 36 visit.
ORG0029 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 5/10/2017, ORG0029 was reportedly hospitalized for a duration of 1 day due to a psychotic episode. We were informed of this information from the participant on 6/8/2017, during their Week 36 visit.
ORG0079 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 5/29/2017, ORG0079 was reportedly hospitalized for a duration of 19 days due to a psychotic episode. We were informed of this information from the participant on 6/22/2017, during their Week 36 visit.
ORG0098 (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) — On 11/25/2016, ORG0098 was reportedly hospitalized for a duration of 12 days due to suicidal thoughts or behaviors. On 3/15/2017, ORG0098 was reportedly hospitalized for a duration of 7 days due to suicidal thoughts or behaviors.
ORG0084 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 1/15/2017, ORG0084 was reportedly hospitalized for a duration of 14 days due to suicidal thoughts or behaviors. We were informed of this information from the participant on 7/13/2017, during their Week 36 visit.
ORG0093 (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — On 2/4/2017, ORG0093 was reportedly hospitalized for a duration of 10 days due to suicidal thoughts or behaviors. We were informed of this information from the participant on 7/18/2017, during their Week 36 visit.
ORG0087 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 4/4/2017, ORG0087 was reportedly hospitalized for a duration of 9 days due to a psychotic episode. We were informed of this information from the participant on 7/19/2017, during their Week 36 visit.
ORG101 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 6/15/2017, ORG0101 was reportedly hospitalized for a duration of 1 day due to suicidal thoughts or behaviors. We were informed of this information from the participant on 7/18/2017, during their Week 36 visit.
ORG0012 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 6/22/2017, ORG0012 was reportedly hospitalized for a duration of 7 days due to a psychotic episode. We were informed of this information from the participant on 10/4/2017, during their Week 52 visit.
ORG0019 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 9/1/2017, ORG0019 was reportedly hospitalized for a duration of 30 days due to a psychotic episode. We were informed of this information from the participant on 10/3/2017, during their Week 52 visit.
ORG0022 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 9/8/2017, ORG0022 was reportedly hospitalized for a duration of 14 days due to suicidal thoughts or behaviors. We were informed of this information from the participant on 10/9/2017, during their Week 52 visit.
ORG0013 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 9/10/2017, ORG0013 was reportedly hospitalized for a duration of 4 days due to "a high anxiety level". We were informed of this information from the participant on 10/5/2017, during their Week 52 visit.
ORG0246 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 9/15/2017, ORG0246 was reportedly hospitalized for a duration of 5 days due to suicidal thoughts or behavior. We were informed of this information from the participant on 3/19/2018, during their Week 36 visit.
ORG0327 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 9/15/2017, ORG0327 was reportedly hospitalized for a duration of 7 days due to a drug or alcohol overdose. We were informed of this information from the participant on 5/22/2018, during their Week 36 visit.
ORG0346 (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — On 10/25/2017, ORG0346 was reportedly hospitalized for a duration of 11 days due to a psychotic episode. On 6/5/2018, ORG0346 was reportedly hospitalized for a duration of 21 days for "drug rehab and depression".
ORG0198 (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — On 10/28/2017, ORG0198 was reportedly hospitalized for a duration of 2 days due to a psychotic episode. We were informed of this information from the participant on 11/14/2017, during their Week 36 visit.
ORG0299 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 1/16/2018, ORG0299 was reportedly hospitalized for a duration of 28 days due to alcohol use. We were informed of this information from the participant on 5/21/2018, during their Week 36 visit.
ORG0162 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 2/2/2018, ORG0162 was reportedly hospitalized for a duration of 7 days due to homicidal or aggressive behavior. We were informed of this information from the participant on 2/12/2018, during their Week 52 visit.
ORG0203 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 4/11/2018, ORG0203 was reportedly hospitalized for a duration of 8 days due to suicidal thoughts or behavior. We were informed of this information from the participant on 6/26/2018, during their Week 52 visit.
ORG0305 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 1/15/2018, ORG0305 was reportedly hospitalized for a duration of 21 days due to a psychotic episode. We were informed of this information from the participant on 9/17/2018, during their Week 52 visit.
ORG0415 (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — On 5/21/2018, ORG0415 was reportedly hospitalized for a duration of 30 days due to an unknown reason. On 5/21/2018, ORG0415 was reportedly hospitalized for a duration of 14 days due to suicidal thoughts or behavior.
ORG0374 (Psychiatric disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) — On 2/15/2018, ORG0374 was reportedly hospitalized for a duration of 6 days due to self-harm. On 9/15/2018, ORG0374 was reportedly hospitalized for a duration of 6 days due to suicidal thoughts or behavior.
ORG0348 (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — On 4/15/2018, ORG0348 was reportedly hospitalized for a duration of 28 days due suicidal thoughts or behavior. On 9/24/2018, ORG0348 was reportedly hospitalized for a duration of 21 day due to a psychotic episode.
ORG0390 (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — On 4/26/2018, ORG0390 was reportedly hospitalized for a duration of 14 days due to suicidal thoughts or behavior. On 6/29/2018, ORG0390 was reportedly hospitalized for a duration of 7 days due to an unknown reason
ORG0426 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 6/13/2018, ORG0426 was reportedly hospitalized for a duration of 1 day due to "medication change". We were informed of this information from the participant on 10/23/2018, during their Week 36 visit.
ORG0362 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 7/15/2018, ORG0362 was reportedly hospitalized for a duration of 21 days due to an unknown reason. We were informed of this information from the participant on 10/16/2018, during their Week 36 visit.
ORG0367 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 8/5/2018, ORG0367 was reportedly hospitalized for a duration of 30 days due to suicidal thoughts or behavior. We were informed of this information from the participant on 2/14/2019, during their Week 52 visit.
ORG0380 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 8/16/2018, ORG0380 was reportedly hospitalized for a duration of 33 days due to a psychotic episode. We were informed of this information from the participant on 10/15/2018, during their Week 36 visit.
ORG0487 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 9/1/2018, ORG0487 was reportedly hospitalized for a duration of 14 days due to a drug or alcohol overdose. We were informed of this information from the participant on 1/8/2019, during their Week 36 visit.
ORG0364 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 9/8/2018, ORG0364 was reportedly hospitalized for a duration of 6 days due to homicidal or aggressive behavior. We were informed of this information from the participant on 10/15/2018, during their Week 36 visit.
ORG0372 (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — On 10/2/2018, ORG0372 was reportedly hospitalized for a duration of 7 days due to suicidal thoughts or behaviors. On 1/15/2019, ORG0372 was reportedly hospitalized for a duration of 7 days due to suicidal thoughts or behaviors.
ORG0421 (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — On 10/10/2018, ORG0421 was reportedly hospitalized for a duration of 5 days due to a psychotic episode. On 11/7/2018, ORG0421 was reportedly hospitalized for a duration of 23 days "to be put on medication".
ORG0389 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 12/25/2018, ORG0389 was reportedly hospitalized for a duration of 5 days due to a psychotic episode. We were informed of this information from the participant on 2/13/2019, during their Week 52 visit.
ORG0425 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On 2/6/2019, ORG0425 was reportedly hospitalized for a duration of 7 days due to "drug rehab". We were informed of this information from the participant on 2/13/2019, during their Week 52 visit.
ORG0475 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 2/27/2019, ORG0475 was reportedly hospitalized for a duration of 28 days due to an unknown reason. We were informed of this information from the participant on 4/17/2019, during their Week 52 visit.
ORG0479 (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On 4/6/2019, ORG0479 was reportedly hospitalized for a duration of 13 days due to a psychotic episode. We were informed of this information from the participant on 4/18/2019, during their Week 52 visit.
ORG0620 (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — they reported they were hospitalized on 12/10/2019 for 30 days for a psychotic episode. they reported they were hospitalized on 9/15/2019 for 2 days for a medication adjustment. They were also hospitalized on 6/15/2019 for 7 days for the same reason.
ORG0705 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — During ORG0705 Week 36 session, they reported they were hospitalized on 9/26/2019 for 9 days for self-harm.
ORG0759 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — During ORG0759 Week 36 session, they reported they were hospitalized on 1/15/2020 for 14 days for a psychotic episode.
ORG0619 (General disorders) | 1 (1) | 0 (0) | NA | NA — On 3/26/2020, we were informed that ORG0619 is in rehab for an unknown duration.
ORG0740 (General disorders) | 1 (1) | 0 (0) | NA | NA — During ORG0740 Week 36 session, they reported they were hospitalized on 7/25/2019 for 16 days for an unknown reason
ORG0727 (Psychiatric disorders) | 1 (1) | 0 (0) | NA | NA — During ORG0727 Week 36 session, they reported they were hospitalized on 12/3/2019 for 14 days for a psychotic episode.
ORG0772 (General disorders) | 1 (1) | 0 (0) | NA | NA — On 05/14/2020, we were informed that ORG0772 was in the hospital due to COVID-19 complications.
ORG0922 (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA — On 11/23/2020, during the ORG0922 baseline session ppt expressed that he had been in the hospital for 12 days problems going to the bathroom.
ORG0881 (General disorders) | 0 (0) | 1 (1) | NA | NA — On 3/18/2021 during the Week 12 session, ORG0881 informed a research team member that they were in the hospital from 2/18/2021-3/10/2021 due to being "302'd" (involuntarily admitted) by their sister and for having Covid-19.
ORG0920 (Social circumstances) | 0 (0) | 1 (1) | NA | NA — On 5/26/2021 during the Week 24 session, ORG0920 reported that she'd been in a car accident on 5/17/21. As of 5/26 she is still in the hospital and cannot walk, but she is getting physical therapy.
ORG0880 (Renal and urinary disorders) | 0 (0) | 1 (1) | NA | NA — On 8/18/2021 ORG0880 reported that she had been hospitalized on 7/24/2021 for a kidney infection. She spent 5 days at the hospital before being transferred to Immaculate Mary for inpatient rehab, which ended on 8/12/2021.
ORG0101 (Psychiatric disorders) | 0 (0) | 1 (1) | NA | NA — On 6/15/2017, ORG0101 was reportedly hospitalized for a duration of 1 day due to suicidal thoughts or behaviors. We were informed of this information from the participant on 7/18/2017, during their Week 36 visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT02849652/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02849652/ICF_000.pdf